CLINICAL TRIAL: NCT00002447
Title: An Open Label, Randomized, Multicenter Study to Evaluate Fortovase (Saquinavir) SGC QD, Norvir (Ritonavir) QD Plus Two NRTIs Vs Sustiva (Efavirenz) QD Plus Two NRTIs in HIV Infected Patients
Brief Title: A Study to Compare Two Anti-HIV Drug Combinations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229R; NR15720C/M61027
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-01

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Saquinavir; HIV Protease Inhibitors; Ritonavir; Dosage Forms; Reverse Transcriptase Inhibitors; Anti-HIV Agents; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; efavirenz; Saquinavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Efavirenz
Drug: Saquinavir

SUMMARY:
The purpose of this study is to compare 2 anti-HIV drug combinations.

DETAILED DESCRIPTION:
Patients are stratified by HIV RNA: 5,000-75,000 vs greater than 75,000 copies/ml by Amplicor assay. Patients are randomized to two arms. Arm A receives SQV plus RTV plus two NRTIs. Arm B receives EFV plus two NRTIs. Patients must take their dose at approximately the same time every day. Patients have the option of taking daily dose in AM or PM. Patients are evaluated for changes in plasma HIV RNA levels and CD4/CD8 counts and for adverse experiences and laboratory determinations. Evaluations are made every 4-8 weeks until Week 48. Patients continuing beyond Week 48 who reach Weeks 60, 72, 84, and common study closure, will be seen at those weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load of at least 5,000 copies/ml and a CD4 cell count of at least 75 cells/mm3.
* Are at least 18.
* Are able to complete the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken any anti-HIV medications for more than 2 weeks.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: JSG Montaner, Principal Investigator; Ann Collier, Study Chair; Danielle Rouleau, Study Chair; Michael Saag, Study Chair; Paul Volberding, Study Chair; Sharon Walmsley, Study Chair; Nicholas Bellos, Study Chair; Alfred Burnside, Study Chair; Stephen Follansbee, Study Chair; Joseph Gathe, Study Chair; Bruce Hathaway, Study Chair; Margaret Hoffman-Terry, Study Chair; Jazila Mantis, Study Chair; Joseph Masci, Study Chair; Mahmoud Mustafa, Study Chair; John Schrank, Study Chair; Malte Schutz, Study Chair; Leon Smith, Study Chair
Locations (26):
- United States (22):
  - Univ of Alabama at Birmingham / AIDS Outpatient Clinic, Birmingham, Alabama
  - St Mary's Med Ctr, Long Beach, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Physicans Home Service, Washington D.C., District of Columbia
  - Associates in Research, Fort Myers, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Illinois Masonic Med Ctr, Chicago, Illinois
  - Saint Michael's Med Ctr / Dept of Infectious Diseases, Newark, New Jersey
  - Infectious Disease Specialists of NJ, Union, New Jersey
  - Elmhurst Hosp, Elmhurst, New York
  - Queens Hospital Center, Jamaica, New York
  - LIJMC, New Hyde Park, New York
  - East Carolina Univ School of Medicine, Greenville, North Carolina
  - Lehigh Valley Hosp, Allentown, Pennsylvania
  - Burnside Clinic, Columbia, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Nicholas Bellos, Dallas, Texas
  - Joseph Gathe, Houston, Texas
  - Univ of Utah, Salt Lake City, Utah
  - Univ of Washington / AIDS Clinical Trial Unit, Seattle, Washington
- Canada (3):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Toronto Gen Hosp, Toronto, Ontario
  - Centre Hospitalier de la Universite de Montreal (CHUM), Montreal, Quebec
- Ponce Univ Hosp, Ponce, Puerto Rico